CLINICAL TRIAL: NCT06566625
Title: The Karolinska Pilot Study for Cardiac Magnetic Resonance Imaging Prior to Invasive Coronary Angiography in Patients With Suspected Non-ST-Elevation Myocardial Infarction
Brief Title: Cardiac MRI Prior to Invasive Coronary Angiography in Patients With Suspected Non-ST-Elevation Myocardial Infarction
Acronym: KaPSICA-CMR
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-02286-01; Dnr 2024-02286-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2024-07-02; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-06

CONDITIONS: Non-ST Elevation Myocardial Infarction; Acute Coronary Syndrome
Keywords: CMR; MRI; Cardiac MRI; Cardiac Magnetic Resonance; Cardiac Magnetic Resonance imaging; AMI; ACS; Acute Coronary Syndrome; NSTEMI; Non-STEMI; ICA; Invasive Coronary Angiography; Coronary Angiography; T1; T2; Magnetic Resonance Fingerprinting; Native T1; Native T2; Magnetic Resonance Angiography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Acute Coronary Syndrome | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: Inclusion criteria:
  ≥18 years of age Suspected NSTEMI (signs and symptoms suggest of ACS with initial ECG showing no ST-elevation) Planned ICA where CMR can be performed without delaying ICA Able to provide written informed consent
  Exclusion criteria:
  Contraindications for CMR examination with gadolinium contrast (claustrophobia, eGFR <30ml/min/1.73m2, contrast allergy, and non-MRI compatible implants) Arrythmias which hinder CMR examination Previous CABG Hemodynamic instability Myocardial infarction <6 months prior to inclusion
  Interventions: Diagnostic Test: Cardiac MRI (CMR) examination

INTERVENTIONS:
Diagnostic Test: Cardiac MRI (CMR) examination — An MRI examination of the heart (CMR) is presently performed as a follow-up examination in patients where an invasive coronary angiography (ICA) shows no obstructive findings. The intervention in this study is characterized by having the CMR performed before, rather than after, the ICA.
  In addition, this study will implement some novel CMR sequences which have not been previously tested in this patient cohort:
  * CMR Angiography (imaging the coronary arteries using MRI)
  * CMR Fingerprinting (sequences which perform T1 and T2 mapping simultaneously)
  Other Names: cmr; cardiac mri; cmr angiography; cmr fingerprinting; fingerprinting; t1 mapping; t2 mapping

SUMMARY:
Patients with a suspected myocardial infarction are subdivided into ST-elevation and non-ST-elevation myocardial infarctions (STEMI and NSTEMI, respectively) using an ECG. While patients with STEMI are urgently referred to a cath lab, patients with NSTEMI usually undergo a planned invasive coronary angiography (ICA) anywhere from 24-72 hours after arriving to the hospital. When an invasive coronary angiography can not explain the cause of a myocardial infarction, an MRI of the heart (a CMR) is often done as a follow-up investigation.

A growing body of evidence suggests that performing a CMR before the planned ICA can provide an accurate diagnosis and defer the need for an ICA in many of these patients with NSTEMI.

DETAILED DESCRIPTION:
KaPSICA-CMR is an observational pilot study at the Karolinska University Hospital which aims to validate, in a Swedish healthcare setting, the potentials of a CMR-first approach in patients with suspected NSTEMI. We plan on including 150 patients, both with (n=50) and without (n=100) previous myocardial infarction. In addition to a standard clinical CMR protocol, the study will test novel CMR techniques such as magnetic resonance angiography and magnetic resonance fingerprinting sequences in this cohort. Patients will be recruited at both the Solna- and Huddinge sites of the hospital and include patients referred to ICA from the Visby- and Södertälje hospitals. The findings on the CMR will be blinded to treating physicians, with exceptions for unexpected adverse findings. In the event that a CMR would be indicated in line with clinical practice, the CMR findings are unblinded.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age Suspected NSTEMI (signs and symptoms suggest of ACS with initial ECG showing no ST-elevation)
* Planned ICA where CMR can be performed without delaying ICA
* Able to provide written informed consent

Exclusion Criteria:

* Contraindications for CMR examination with gadolinium contrast (claustrophobia, eGFR <30ml/min/1.73m2, contrast allergy, and non-MRI compatible implants)
* Arrythmias which hinder CMR examination
* Previous CABG
* Hemodynamic instability
* Myocardial infarction <6 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present with suspected NSTEMI and have a planned invasive coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of non-ischemic diagnosis | Every three months, until study completion
  In cases where CMR establishes a diagnosis which is non-ischemic in nature, such as a myocarditis, an ICA can be deferred since a diagnosis has been made using CMR.
Rate of IRA territory reclassification | Every three months, until study completion
  One primary outcome measurement will be to what extent a CMR examination can reclassify the IRA (infarct-related artery) territory established on ICA, by designating a new IRA based on the area of infarction on CMR using the 17-segment model of the American Heart Association and magnetic resonance angiography

CONTACTS AND LOCATIONS:
Overall Officials: Marcus E Carlsson, Professor, Principal Investigator — Karolinska Insitutet and Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden